CLINICAL TRIAL: NCT05296824
Title: Cryoballoon Isolation of Combined Posterior Wall and Pulmonary Veins Versus Pulmonary Veins Alone for the Treatment of Paroxysmal Atrial Fibrillation (IMPPROVE-PAF)
Brief Title: Cryoballoon PVI With PWI Versus PVI Alone In Patients With PAF
Status: Completed | Type: Observational
Sponsor: Sacramento EP Research (Other)
Collaborators: Mercy General Hospital and Dignity Health Heart and Vascular Institute (Unknown); UC Health Medical Center (Unknown); The University of Texas Health Science Center, Houston (Other); Beth Israel Deaconess Medical Center (Other)
Responsible Party: Principal Investigator, Arash Aryana, MD, Director, Greater Sacramento Cardiovascular Service Line, Sacramento EP Research
Other Study IDs: IMPPROVE-PAF
Record Dates: First submitted 2022-03-16; First posted 2022-03-25 (Actual); Results first posted 2025-11-05 (Actual); Last update posted 2025-11-05 (Actual); Status verified 2025-10

CONDITIONS: Paroxysmal Atrial Fibrillation
Keywords: Cryoballoon; Pulmonary vein isolation; Posterior wall isolation; Paroxysmal atrial fibrillation
MeSH Terms: conditions — Atrial Fibrillation

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (2):
- Pulmonary vein isolation (PVI) only: Patients with symptomatic paroxysmal atrial fibrillation who received cryoballoon pulmonary vein isolation (PVI) only
  Interventions: Procedure: Cryoballoon ablation for the treatment of atrial fibrillation
- Pulmonary vein isolation (PVI) with posterior wall isolation (PWI): Patients with symptomatic paroxysmal atrial fibrillation who received cryoballoon pulmonary vein isolation (PVI) with posterior wall isolation (PWI)
  Interventions: Procedure: Cryoballoon ablation for the treatment of atrial fibrillation

INTERVENTIONS:
Procedure: Cryoballoon ablation for the treatment of atrial fibrillation — Cryoballoon ablation for the treatment of atrial fibrillation

SUMMARY:
Cryoballoon ablation has emerged as a safe and effective strategy for treatment of atrial fibrillation (AF) for which it has recently received a 'first-line' therapy indication by the FDA. Pulmonary vein (PV) isolation (PVI) has been the cornerstone of this procedure achieving freedom from recurrent AF in up to ~80% of patients at 12 months of follow-up. However, the success has been shown to be significantly lower, in the range of 50-60% at 3-5 years of follow-up. Other more recent cryoballoon ablation studies have demonstrated marked improvements in clinical outcomes associated with concomitant PVI and cryoballoon ablation/isolation of the 'PV component' (a region of the left atrial posterior [back] wall lying between the PVs that is anatomically and embryologically related to the PVs), versus PVI alone in patients with persistent AF.

PVI+PWI using cryoballoon ablation has been widely-practiced in patients with paroxysmal AF. However, the acute/long-term safety and efficacy of this approach has not been formally investigated in paroxysmal AF. Given the mechanistic similarities between persistent and paroxysmal AF, the investigators hypothesize that similar benefits associated with PVI+PWI may also be observed in those with paroxysmal AF. Yet, due to the relative infrequency of breakthrough/recurrent arrhythmias in patients with PAF, to detect a significant difference, large sample sizes and extended follow-up (>24 months) are likely needed. Hence, the aim of this retrospective, observational study is to examine the acute and long-term efficacy and safety beyond 36 months of follow-up associated with PVI alone versus PVI+PWI using cryoballoon ablation in a large cohort of patients with PAF, performed by a single operator between 1/1/2014 and 8/31/2018 at Mercy General Hospital.

DETAILED DESCRIPTION:
INTRODUCTION AND RATIONALE Cryoballoon ablation has emerged as a safe and effective strategy for the treatment of atrial fibrillation (AF), and based on growing evidence, it recently received an initial rhythm control strategy ('first-line' therapy) indication by the Food and Drug Administration. Pulmonary vein (PV) isolation (PVI) guided typically by cryoballoon PV occlusion remains the cornerstone of cryoballoon ablation. Although single-procedure freedom from recurrent AF following such an approach has been reported to be as high as 82% at 12 months, the success appears to be markedly diminished in the range of 50-60% during long-term follow-up. This in part may be related to the inherent limitations of cryoballoon ablation which often yields an ostial (distal) level PVI. Along these lines, prior investigations have found wide-area antral PVI encompassing the PV component (i.e., the region of the posterior wall lying between the PVs) to be superior to ostial PVI. Other more recent studies involving the cryoballoon have demonstrated marked improvements in clinical efficacy associated with concomitant PVI and posterior wall isolation (PWI) within the region of the PV component as compared to PVI alone, in patients with persistent AF. Though widely-practiced, this approach has not been formally investigated in patients with symptomatic paroxysmal AF (PAF). Given the mechanistic similarities between persistent and PAF, the investigators hypothesize that similar benefits may also be observed with PVI+PWI in the patients with PAF. Yet, given the relative infrequency of breakthrough/recurrent arrhythmias in patients with PAF, to detect a significant difference, large sample sizes and extended follow-up (>24 months) are likely needed. Hence, the aim of this retrospective, observational study is to examine the clinical efficacy and safety of PVI alone versus PVI+PWI using cryoballoon ablation, in a large cohort of patients with symptomatic PAF beyond 36 months of follow-up.

EMBRYOLOGIC EVIDENCE The PV component of the posterior left atrial wall shares a common primordial origin with the PVs. The embryologic origin of the four PVs and the PV component can be traced back to the mediastinal myocardium derived from a mid-pharyngeal strand at 6 weeks of gestation. Early on during development, a single primitive vein returns blood from the lungs to the common trabeculated atrium. As the interatrial septum forms, the single vein divides twice to give rise to the four PVs. As the PV ostia migrate away from one another, the smooth tissue of the posterior left atrial wall forms. Although this region is anatomically contiguous with the surrounding trabeculated tissue from the primitive left atrium, its embryologic origin results in electrophysiologic properties that are more similar to the muscular PV sleeves than the immediately adjacent atrial roof or floor ('true' posterior wall).

During embryogenesis, the single vein and its surrounding tissue (in addition to the Bachmann's bundle and sinus venosus-derived structures) demonstrate the expression of genes responsible for development of cardiac conduction system. Although expression of these genes decreases during embryogenesis, it is hypothesized that their continued low-level expression may explain why certain regions within the atria are more commonly the site of origin of focal ectopy. These embryologic characteristics would certainly explain the well-accepted clinical observation that AF is frequently initiated by ectopic beats arising from the PVs and the increasingly reported observation that ectopic beats from the left atrial posterior wall can similarly initiate AF.

ANATOMIC EVIDENCE A visual examination of the PV component and the orientation of its myofibrils suggests direct continuity between this region and the PV antra as does a gross anatomical assessment of certain left atrial morphologies. Meanwhile, underneath the smooth endocardial surface of the PV component, numerous subendocardial and subepicardial muscular bundles traverse with varying fiber orientation. Fibers immediately surrounding the PVs typically encircle the veins, whereas those in the subepicardial aspect of the posterior wall are comprised of the septo-pulmonary bundle and display a more vertical or oblique orientation. Immediately adjacent to the lateral aspect of the septo-pulmonary bundle are found transversely oriented fibers which extend to the left PV ostia. It is this change in orientation that is believed to promote anisotropic conduction and therefore reentry.

Prior investigators have found that in patients with PAF, this juxtaposition of fiber orientations was associated with isochronal crowding and functional block depending on the direction of wave front propagation during sinus or paced rhythm. Similarly, mapping of fibrillatory waves during cardiac surgery in patients with AF has revealed simultaneous propagation of longitudinally dissociated fibrillation waves which are separated by continuously changing lines of block. These lines of block are once again most densely packed in the PV component, leading to the highest degree of block and dissociation and the lowest incidence of wave front boundaries formed by collision.

ELECTROPHYSIOLOGIC EVIDENCE As discussed, the PV component is derived from tissues other than the primitive cardiac tube. Hence, the PV component is believed to be related more to PV versus atrial tissue. Some studies have suggested that these tissues share more in common with the sinoatrial nodal myocytes, displaying higher diastolic calcium contents and propensity to spontaneous depolarization. Furthermore, the PV component exhibits increased conduction abnormalities, a higher incidence of delayed after depolarizations and larger late sodium and intracellular and sarcoplasmic reticulum Ca++ contents, but a smaller inward rectifier potassium currents and a reduced resting membrane potential. The posterior wall and the PV myocytes are also characterized by shorter action potential durations and slower phase 0 upstroke velocities. As such, the PV component is believed to be the site of collision of activation wave fronts as they sweep across the left atrial dome. Along these lines, prior Investigators have found this region of the left atrium to be responsible for 80% of high-frequency rotors in an isolated sheep heart model. Similarly, mapping in humans often localizes stable rotors or focal sources as well as complex fractionated electrograms in the posterior wall and the left atrial roof. The PV component has in fact been shown to be a common source of triggers accounting for up to ~40% of non-PV triggers in patients with AF.

Lastly, the PV component is also the site of the main autonomic ganglionic plexi related to the left atrial dome (i.e., the superior left atrial ganglionated plexus) which is believed to modulate extrinsic cardiac innervation and facilitate the occurrence of AF in a hyperactive autonomic state. As such, it is believed that catheter ablation of the PV component also greatly attenuates the input of these plexi to the PVs, interrupting the vagosympathetic input to the ligament of Marshall and the inferior left ganglionated plexus which have been highly implicated in the pathogenesis of AF.

ELIGIBILITY:
Inclusion Criteria:

* Age 18 years or older
* Cryoballoon PVI+PWI
* Cryoballoon PVI alone
* Symptomatic paroxysmal atrial fibrillation

Exclusion Criteria:

* None

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Patients with symptomatic paroxysmal atrial fibrillation
Sampling Method: Probability Sample
Enrollment: 320 (Actual)
Dates: Start 2014-01-01 (Actual); Primary Completion 2018-08-31 (Actual); Study Completion 2021-12-31 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Arash Aryana, MD, PhD, Principal Investigator — Mercy General Hospital and Dignity Health Heart and Vascular Institute
Locations (4):
- United States (4):
  - Mercy General Hospital and Dignity Health Heart and Vascular Institute, Sacramento, California
  - UC Health Medical Center, Loveland, Colorado
  - Beth Israel Deaconess Medical Center, Boston, Massachusetts
  - University of Texas Health Science Center at Houston, Houston, Texas

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Haissaguerre M, Jais P, Shah DC, Takahashi A, Hocini M, Quiniou G, Garrigue S, Le Mouroux A, Le Metayer P, Clementy J. Spontaneous initiation of atrial fibrillation by ectopic beats originating in the pulmonary veins. N Engl J Med. 1998 Sep 3;339(10):659-66. doi: 10.1056/NEJM199809033391003. PMID 9725923
- [Background] Kuniss M, Pavlovic N, Velagic V, Hermida JS, Healey S, Arena G, Badenco N, Meyer C, Chen J, Iacopino S, Anselme F, Packer DL, Pitschner HF, Asmundis C, Willems S, Di Piazza F, Becker D, Chierchia GB; Cryo-FIRST Investigators. Cryoballoon ablation vs. antiarrhythmic drugs: first-line therapy for patients with paroxysmal atrial fibrillation. Europace. 2021 Jul 18;23(7):1033-1041. doi: 10.1093/europace/euab029. PMID 33728429
- [Background] Aryana A, Kenigsberg DN, Kowalski M, Koo CH, Lim HW, O'Neill PG, Bowers MR, Hokanson RB, Ellenbogen KA; Cryo-DOSING Investigators. Verification of a novel atrial fibrillation cryoablation dosing algorithm guided by time-to-pulmonary vein isolation: Results from the Cryo-DOSING Study (Cryoballoon-ablation DOSING Based on the Assessment of Time-to-Effect and Pulmonary Vein Isolation Guidance). Heart Rhythm. 2017 Sep;14(9):1319-1325. doi: 10.1016/j.hrthm.2017.06.020. Epub 2017 Jun 15. PMID 28625929
- [Background] Kis Z, Muka T, Franco OH, Bramer WM, De Vries LJ, Kardos A, Szili-Torok T. The Short and Long-Term Efficacy of Pulmonary Vein Isolation as a Sole Treatment Strategy for Paroxysmal Atrial Fibrillation: A Systematic Review and Meta-Analysis. Curr Cardiol Rev. 2017;13(3):199-208. doi: 10.2174/1573403X13666170117125124. PMID 28124593
- [Background] Reddy VY, Neuzil P, d'Avila A, Laragy M, Malchano ZJ, Kralovec S, Kim SJ, Ruskin JN. Balloon catheter ablation to treat paroxysmal atrial fibrillation: what is the level of pulmonary venous isolation? Heart Rhythm. 2008 Mar;5(3):353-60. doi: 10.1016/j.hrthm.2007.11.006. Epub 2007 Nov 7. PMID 18313591
- [Background] Mesquita J, Cavaco D, Ferreira AM, Costa FM, Carmo P, Morgado F, Mendes M, Adragao P. Very long-term outcomes after a single catheter ablation procedure for the treatment of atrial fibrillation-the protective role of antiarrhythmic drug therapy. J Interv Card Electrophysiol. 2018 Jun;52(1):39-45. doi: 10.1007/s10840-018-0340-4. Epub 2018 Mar 6. PMID 29511973
- [Background] McLellan AJ, Ling LH, Azzopardi S, Lee GA, Lee G, Kumar S, Wong MC, Walters TE, Lee JM, Looi KL, Halloran K, Stiles MK, Lever NA, Fynn SP, Heck PM, Sanders P, Morton JB, Kalman JM, Kistler PM. A minimal or maximal ablation strategy to achieve pulmonary vein isolation for paroxysmal atrial fibrillation: a prospective multi-centre randomized controlled trial (the Minimax study). Eur Heart J. 2015 Jul 21;36(28):1812-21. doi: 10.1093/eurheartj/ehv139. Epub 2015 Apr 28. PMID 25920401
- [Background] Reissmann B, Budelmann T, Wissner E, Schluter M, Heeger CH, Mathew S, Maurer T, Lemes C, Fink T, Rillig A, Santoro F, Riedl J, Ouyang F, Kuck KH, Metzner A. Five-year clinical outcomes of visually guided laser balloon pulmonary vein isolation for the treatment of paroxysmal atrial fibrillation. Clin Res Cardiol. 2018 May;107(5):405-412. doi: 10.1007/s00392-017-1199-6. Epub 2017 Dec 28. PMID 29285621
- [Background] Aryana A, Baker JH, Espinosa Ginic MA, Pujara DK, Bowers MR, O'Neill PG, Ellenbogen KA, Di Biase L, d'Avila A, Natale A. Posterior wall isolation using the cryoballoon in conjunction with pulmonary vein ablation is superior to pulmonary vein isolation alone in patients with persistent atrial fibrillation: A multicenter experience. Heart Rhythm. 2018 Aug;15(8):1121-1129. doi: 10.1016/j.hrthm.2018.05.014. PMID 30060879
- [Background] Elbatran AI, Anderson RH, Mori S, Saba MM. The rationale for isolation of the left atrial pulmonary venous component to control atrial fibrillation: A review article. Heart Rhythm. 2019 Sep;16(9):1392-1398. doi: 10.1016/j.hrthm.2019.03.012. Epub 2019 Mar 16. PMID 30885736
- [Background] Clarke JD, Piccini JP, Friedman DJ. The role of posterior wall isolation in catheter ablation of persistent atrial fibrillation. J Cardiovasc Electrophysiol. 2021 Sep;32(9):2567-2576. doi: 10.1111/jce.15164. Epub 2021 Jul 21. PMID 34258794
- [Background] Aryana A, Su W, Kuniss M, Okishige K, de Asmundis C, Tondo C, Chierchia GB. Segmental nonocclusive cryoballoon ablation of pulmonary veins and extrapulmonary vein structures: Best practices III. Heart Rhythm. 2021 Aug;18(8):1435-1444. doi: 10.1016/j.hrthm.2021.04.020. Epub 2021 Apr 24. PMID 33905811
- [Background] Bisignani A, Overeinder I, Kazawa S, Iacopino S, Cecchini F, Miraglia V, Osorio TG, Boveda S, Bala G, Mugnai G, Monaco C, Stroker E, Brugada P, Sieira J, Galli A, de Asmundis C, Chierchia GB. Posterior box isolation as an adjunctive ablation strategy with the second-generation cryoballoon for paroxysmal atrial fibrillation: a comparison with standard cryoballoon pulmonary vein isolation. J Interv Card Electrophysiol. 2021 Aug;61(2):313-319. doi: 10.1007/s10840-020-00812-z. Epub 2020 Jul 6. PMID 32632544
- [Background] Mun HS, Joung B, Shim J, Hwang HJ, Kim JY, Lee MH, Pak HN. Does additional linear ablation after circumferential pulmonary vein isolation improve clinical outcome in patients with paroxysmal atrial fibrillation? Prospective randomised study. Heart. 2012 Mar;98(6):480-4. doi: 10.1136/heartjnl-2011-301107. Epub 2012 Jan 27. PMID 22285969
- [Background] Kim TH, Park J, Park JK, Uhm JS, Joung B, Hwang C, Lee MH, Pak HN. Linear ablation in addition to circumferential pulmonary vein isolation (Dallas lesion set) does not improve clinical outcome in patients with paroxysmal atrial fibrillation: a prospective randomized study. Europace. 2015 Mar;17(3):388-95. doi: 10.1093/europace/euu245. Epub 2014 Oct 21. PMID 25336665
- [Background] Hindricks G, Piorkowski C, Tanner H, Kobza R, Gerds-Li JH, Carbucicchio C, Kottkamp H. Perception of atrial fibrillation before and after radiofrequency catheter ablation: relevance of asymptomatic arrhythmia recurrence. Circulation. 2005 Jul 19;112(3):307-13. doi: 10.1161/CIRCULATIONAHA.104.518837. Epub 2005 Jul 11. PMID 16009793
- [Background] Mohanty S, Trivedi C, Horton P, Della Rocca DG, Gianni C, MacDonald B, Mayedo A, Sanchez J, Gallinghouse GJ, Al-Ahmad A, Horton RP, Burkhardt JD, Dello Russo A, Casella M, Tondo C, Themistoclakis S, Forleo G, Di Biase L, Natale A. Natural History of Arrhythmia After Successful Isolation of Pulmonary Veins, Left Atrial Posterior Wall, and Superior Vena Cava in Patients With Paroxysmal Atrial Fibrillation: A Multi-Center Experience. J Am Heart Assoc. 2021 Jun;10(11):e020563. doi: 10.1161/JAHA.120.020563. Epub 2021 May 17. PMID 33998277
- [Background] Jalife J, Kaur K. Atrial remodeling, fibrosis, and atrial fibrillation. Trends Cardiovasc Med. 2015 Aug;25(6):475-84. doi: 10.1016/j.tcm.2014.12.015. Epub 2014 Dec 31. PMID 25661032
- [Background] Atienza F, Almendral J, Moreno J, Vaidyanathan R, Talkachou A, Kalifa J, Arenal A, Villacastin JP, Torrecilla EG, Sanchez A, Ploutz-Snyder R, Jalife J, Berenfeld O. Activation of inward rectifier potassium channels accelerates atrial fibrillation in humans: evidence for a reentrant mechanism. Circulation. 2006 Dec 5;114(23):2434-42. doi: 10.1161/CIRCULATIONAHA.106.633735. Epub 2006 Nov 13. PMID 17101853
- [Background] Aryana A, Allen SL, Pujara DK, Bowers MR, O'Neill PG, Yamauchi Y, Shigeta T, Vierra EC, Okishige K, Natale A. Concomitant Pulmonary Vein and Posterior Wall Isolation Using Cryoballoon With Adjunct Radiofrequency in Persistent Atrial Fibrillation. JACC Clin Electrophysiol. 2021 Feb;7(2):187-196. doi: 10.1016/j.jacep.2020.08.016. Epub 2020 Oct 28. PMID 33602399
- [Derived] Aryana A, Thiemann AM, Pujara DK, Cossette LL, Allen SL, Bowers MR, Gandhavadi M, Heath R, Trivedi AD, O'Neill PG, Ellis ER, d'Avila A. Pulmonary Vein Isolation With and Without Posterior Wall Isolation in Paroxysmal Atrial Fibrillation: IMPPROVE-PAF Trial. JACC Clin Electrophysiol. 2023 May;9(5):628-637. doi: 10.1016/j.jacep.2023.01.014. Epub 2023 Mar 22. PMID 37225309

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Consecutive patients with an age greater than 18 years and symptomatic paroxysmal atrial fibrillation who underwent first-time cryoballoon ablation using either pulmonary vein isolation (PVI) alone or pulmonary vein isolation + Posterior Wall Isolation (PVI+PWI) with at least 36 months of follow-up by a single operator between 1/2014 and 12/2018 at Mercy General Hospital, will be included in this retrospective, non-randomized study.
Period: Overall Study
Arm/Group | Pulmonary Vein Isolation (PVI) Only | Pulmonary Vein Isolation (PVI) With Posterior Wall Isolation (PWI)
Started | 160 | 160
Completed | 160 | 160
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Pulmonary Vein Isolation (PVI) Only | Pulmonary Vein Isolation (PVI) With Posterior Wall Isolation (PWI) | Total
Number analyzed (Participants) | 160 | 160 | 320
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 91 | 109 | 200
  >=65 years | 69 | 51 | 120
Age, Continuous [Mean (Standard Deviation); unit: years] | 63 (11) | 63 (10) | 63 (11)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 54 | 61 | 115
  Male | 106 | 99 | 205
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Number; unit: participants]
  United States | 160 | 160 | 320
Symptomatic paroxysmal atrial fibrillation [Count of Participants; unit: Participants] | 160 | 160 | 320

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Recurrent Atrial Fibrillation
Description: The recurrence of atrial fibrillation following PVI+PWI versus PVI alone using cryoballoon ablation in patients with symptomatic paroxysmal atrial fibrillation during long-term follow-up greater than 3 years.
Time Frame: 56 months
Measure: Count of Participants; unit: Participants
Arm/Group | Pulmonary Vein Isolation (PVI) Only | Pulmonary Vein Isolation (PVI) With Posterior Wall Isolation (PWI)
Number analyzed (Participants) | 160 | 160
Participants | 60 | 31

2. Secondary Outcome: Number of Participants With Recurrence of All Atrial Arrhythmias
Description: The recurrence of all atrial arrhythmias following PVI+PWI versus PVI alone using cryoballoon ablation in patients with symptomatic paroxysmal atrial fibrillation during long-term follow-up greater than 3 years.
Time Frame: 56 months
Measure: Count of Participants; unit: Participants
Arm/Group | Pulmonary Vein Isolation (PVI) Only | Pulmonary Vein Isolation (PVI) With Posterior Wall Isolation (PWI)
Number analyzed (Participants) | 160 | 160
Participants | 70 | 36

ADVERSE EVENTS:
Time Frame: 36 months
Description: All subjects' electronic medical records were reviewed for any adverse events or serious adverse events for the 36 month time period following the index ablation.
Arm/Group | Pulmonary Vein Isolation (PVI) Only | Pulmonary Vein Isolation (PVI) With Posterior Wall Isolation (PWI)
All-Cause Mortality (participants affected / at risk) | 0/160 | 0/160
Serious Adverse Events (participants affected / at risk) | 6/160 | 4/160
Other Adverse Events (participants affected / at risk) | 0/160 | 0/160
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Pulmonary Vein Isolation (PVI) Only (N=160) | Pulmonary Vein Isolation (PVI) With Posterior Wall Isolation (PWI) (N=160)
Transient Phrenic Nerve Palsy (Cardiac disorders) | 3 (3) | 1 (1)
Persistent Phrenic Nerve Palsy (Cardiac disorders) | 1 (1) | 0 (0)
Pericardial Effusion (Cardiac disorders) | 2 (2) | 1 (1)
Groin Vascular Complication (Vascular disorders) | 1 (1) | 2 (2)

LIMITATIONS AND CAVEATS:
Nonrandomized analysis despite extensive cohort matching may have confounded either treatment arm; PVI used during initial study phase & later PVI+PWI was used; Follow-up ambulatory ECG monitoring may have failed to detect asymptomatic atrial arrhythmia recurrences; use of implantable cardiac devices vs continuous monitoring; Asymptomatic expressions of certain complications (e.g., esophageal lesions or PV stenosis) could not be entirely excluded as routine diagnostic tests were not performed.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2021-08-08): https://cdn.clinicaltrials.gov/large-docs/24/NCT05296824/Prot_SAP_000.pdf